CLINICAL TRIAL: NCT06434896
Title: Circulating Tumor DNA Based Adjuvant Chemotherapy in Stage II Colon Cancer Patients: the MEDOCC-CrEATE Trial
Acronym: CrEATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Personal Genome Diagnostics (Industry); The Netherlands Cancer Institute (Other)
Responsible Party: Principal Investigator, Miriam Koopman, Prof. dr., UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL71881.041.19
Record Dates: First submitted 2024-04-29; First posted 2024-05-30 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Circulating Tumor DNA; Recurrence; Colon Cancer Stage II
MeSH Terms: conditions — Recurrence; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ctDNA-based treatment group (Experimental): Patients randomized to the ctDNA-based treatment group will have their post-surgery samples analysed directly after informed consent for MEDOCC-CrEATE. Results are reported to the treating physician and patients. All patients with detectable ctDNA are considered high risk stage 2 patients and will be offered adjuvant chemotherapy for 3 months (4 cycles CAPOX) according to routine clinical practice. Patients with undetectable ctDNA will receive routine follow-up at the surgical department.
  Interventions: Other: ctDNA analysis after surgery
- Standard of care group (No Intervention): The treating physician and patient are not informed about the ctDNA result and these patients will receive routine follow-up at the surgical department.

INTERVENTIONS:
Other: ctDNA analysis after surgery — ctDNA analysis of post-surgery blood samples will be performed directly after informed consent for MEDOCC-CrEATE.
  Arms: ctDNA-based treatment group

SUMMARY:
Patients in the Prospective Dutch ColoRectal Cancer cohort (PLCRC) with non-metastatic colon cancer that gave consent for additional blood withdrawals are enrolled in the observational PLCRC-MEDOCC substudy. In this study, blood is collected before surgery, after surgery and during follow-up. Within PLCRC-MEDOCC, patients with stage II colon cancer that are not considered to have an indication for adjuvant chemotherapy, can be included in the MEDOCC-CrEATE subcohort under the condition that they gave informed consent in PLCRC for biobanking of tissue and for future studies (Trial within Cohorts design).

Patients included in MEDOCC-CrEATE will be randomized 1:1 to the (A) ctDNA-based treatment group versus (B) the standard of care group. A total of 1320 patients will be randomized. Patients randomized to the ctDNA-based treatment group will have their post-surgery samples analysed directly after informed consent for MEDOCC-CrEATE. All patients with detectable ctDNA will be offered adjuvant chemotherapy (3 months CAPOX). Patients with undetectable ctDNA will receive routine follow-up at the surgical department. The aim of this Trial within Cohorts study is to investigate how many patients with detectable ctDNA after surgery start with adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Informed consent for PLCRC with specific consent for:

  * additional blood withdrawals
  * collection and use of tissue for scientific research
  * invitation for future (experimental) research within the cohort, including TwiCs studies
* Inclusion in observational PLCRC -MEDOCC substudy
* Histological confirmed stage II colon cancer
* Fit enough to receive treatment with combination chemotherapy (fluoropyrimidine and oxaliplatin) according to the treating physician

Exclusion Criteria:

* Indication for adjuvant chemotherapy according to treating physician
* Another malignancy in previous 5 years, with the exception of treated carcinoma in situ or skin cancer other than melanoma
* Incomplete primary tumor resection (R1 or R2 resection)
* Contra-indication for fluoropyrimidines or oxaliplatin
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1320 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2035-03 (Estimated); Study Completion 2035-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients starting with adjuvant chemotherapy after detection of ctDNA in their blood. | 8-12 weeks after surgery

SECONDARY OUTCOMES:
Recurrence Rate | 2 and 5 years after surgery
  Proportion of patients that will experience disease recurrence
Disease Free Survival rate | 2 and 5 years after surgery
  Proportion of patients that are alive and free of disease
Disease-related Overall Survival rate | 5 years after surgery
  Proportion of patients that are alive
Time to Recurrence | From date of randomization until the date of recurrence, assessed up to 5 years.
Quality of Life after treatment | 10 years
  Quality of Life (QoL) will be measured using questionnaires that are provided to patients who have given informed consent for the collection of questionnaires within PLCRC.
  Comparison of QoL of the ctDNA positive patients in both study arms will be done using repeated measurements methods, including ACT as factor. QoL will also be analysed for the whole population in both arms of the study. Treatment differences at each QoL assessment time point will be compared by means of the Wilcoxon Rank Sum Test.
Cost-effectiveness of the ctDNA-based treatment | 5 years after diagnosis
  The cost-effectiveness analysis will be carried out from a societal perspective, including both direct health care costs as well as indirect costs from productivity loss. The health outcome measure in the cost-effectiveness analysis will be the total quality adjusted life years (QALY) per group.

CONTACTS AND LOCATIONS:
Locations (29):
- Netherlands (29):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuisgroep Twente, Almelo
  - Flevoziekenhuis, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - NKI-AVL, Amsterdam
  - Rijnstate, Arnhem
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Albert Schweizer Ziekenhuis, Dordrecht
  - Ziekenhuis Gelderse Vallei, Ede
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Rivas, Gorinchem
  - Spaarne Gasthuis, Haarlem
  - Ziekenhuis St. Jansdal, Harderwijk
  - Maastricht UMC, Maastricht
  - Van Weel-Bethesda Ziekenhuis, Middelharnis
  - St. Antonius Ziekenhuis, Nieuwegein
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Bravis Ziekenhuis, Roosendaal
  - Ikazia Ziekenhuis, Rotterdam
  - Haaglanden MC, The Hague
  - Bernhoven, Uden
  - Diakonessenhuis, Utrecht
  - UMC Utrecht, Utrecht
  - Maxima Medisch Centrum, Veldhoven
  - VieCuri Medisch Centrum, Venlo
  - St. Jans Gasthuis, Weert